CLINICAL TRIAL: NCT05404867
Title: Study of Structural and Functional Brain Connectivity Changes in ALS (CoALS-II)
Acronym: CoALS-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY02001218
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Functional Magnetic Resonance Imaging; Connectivity; Diffusion Tensor Imaging; Dynamometer
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALS patients (Other): Patients with ALS
  Interventions: Other: fMRI
- Healthy controls (Other): Age-matched healthy controls
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — fMRI scan for 1 hour

SUMMARY:
This study will try to understand the difference in brain structure between ALS patients and healthy people of similar age. ALS is a condition affecting the nervous system with disruption of the brain networks. This study aims to understand these disruptions and determine their significance in ALS.

DETAILED DESCRIPTION:
Participants and healthy controls will be consented into the study. After consent, details including age, duration of disease, ALSFRS score, and grip strength will be collected. Participants will be trained to perform a grip and release task using a foam ball for 1 minute while inside an MRI scanner. Anatomical, functional and diffusion MRI sequences will be acquired during the scanning, and total scan time will be approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Based on El Escorial Criteria we will select Probable or Definite ALS.
* Healthy controls age matched to ALS patients
* Subjects should be able to lie down in a scanner and undergo an hour-long MRI study
* Subjects should be able to understand instructions, provide consent and perform a hand task while inside the scanner

Exclusion Criteria:

* Unable to undergo MRI due to any reason
* Age <18
* ALS patients having high aspiration risk
* Patients having cognitive limitations which prevents them from understanding the study requirements, providing consent or perform tasks inside the scanner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
fMRI | 1 hour
  Brain network generation and analysis will be performed for anatomical and functional imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States